CLINICAL TRIAL: NCT00843687
Title: Comparative Single-Dose Pharmacokinetics and Safety of Gluteal and Deltoid Intramuscular Injection of Long-Acting Injectable Risperidone in Subjects With Chronic Stable Schizophrenia
Brief Title: A Comparison of the Pharmacokinetics and Safety of Long-acting Injectable Risperidone When Administered to Gluteal or Deltoid Intramuscular Injection Sites in Stable Schizophrenia Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR011023
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Long-acting injectable; Intramuscular injection; Pharmacokinetics
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: Risperidone long-acting injectable

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and safety of long-acting injectable risperidone, an atypical antipsychotic medication used for the treatment of patients with schizophrenia, when it is administered as an intramuscular injection via the deltoid muscle, compared with intramuscular injection via the gluteal muscle.

DETAILED DESCRIPTION:
This is a randomized, open label, single dose, multicenter, 2-way crossover study comprising a screening phase, 2 open-label treatment periods, and end-of-study evaluations. The study population will comprise patients with chronic stable schizophrenia. Patients will be allowed to continue on their existing oral antipsychotic treatment throughout the study, if not receiving disallowed mediations, per protocol. Patients will be randomly allocated to receive treatment in 1 of 2 panels. In each panel, patients will receive a single intramuscular injection of long-acting injectable risperidone in each treatment period, in a 2-way crossover design. In Panel I, patients will receive 25 mg long-acting injectable risperidone via the gluteal muscle and 37.5 mg long-acting injectable risperidone via the deltoid muscle during the study period. In Panel II, patients will receive 50 mg long-acting injectable risperidone via the gluteal muscle and 50 mg long-acting injectable risperidone via the deltoid muscle. There will be a washout period of 85 days between each administration of study drug. The primary outcome will be comparison of the pharmacokinetic parameters area under the curve (AUC) and peak plasma concentration (Cmax) for 37.5 mg deltoid versus 25 mg gluteal, and for 50 mg deltoid versus 50 mg gluteal. Safety will be assessed at screening, throughout the open-label treatment phase, and at the end of study or early withdrawal using a combination of adverse events (including occurrence of extrapyramidal symptoms as assessed by the Extrapyramidal Symptoms Rating Scale), clinical laboratory tests (hematology, serum chemistry, urinalysis, and pregnancy testing), vital signs, physical examinations, electrocardiograms, and injection site evaluation. The study hypothesis is that intramuscular injections of long-acting injectable risperidone via the gluteal and deltoid sites will be bioequivalent routes of administration, as measured by peak and total drug concentrations in the plasma, and that the safety and tolerability profiles of the 2 injection sites will be comparable. The patients will receive a single injection of long--acting injectable risperidone (25 mg, 37.5 mg or 50 mg) in their gluteal or deltoid muscle in 2 treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Chronic schizophrenia of any subtype, according to Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV) criteria
* stable schizophrenia without any changes in medications or dosage during the 4 weeks before the screening visit
* Clinical Global Impression scale score of <=3 (mild)
* informed consent signed by the patient
* patient is otherwise healthy on the basis of a prestudy physical examination and medical history.

Exclusion Criteria:

* No DSM-IV Axis I diagnosis other than schizophrenia
* no pregnant or breast feeding women
* no female subject of childbearing potential without adequate contraception
* no history of severe drug allergy or hypersensitivity
* no patients with inadequate mass in the gluteal or deltoid regions to receive the intramuscular drug injections.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2005-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Comparison of the pharmacokinetic parameters AUC and Cmax for 37.5 mg deltoid versus 25 mg gluteal, and for 50 mg deltoid versus 50 mg gluteal based on blood sampling at predefined intervals up to 85 days.

SECONDARY OUTCOMES:
Patient-rated local site injection pain (measured on a visual analogue scale) & investigator-rated local site injection reaction (measured by injection site evaluation scale) measured 30 min. before injection & at regular intervals up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A comparison of the pharmacokinetics and safety of long-acting injectable risperidone when administered to gluteal or deltoid intramuscular injection sites in stable schizophrenia patients. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=724&filename=CR011023_CSR.pdf